CLINICAL TRIAL: NCT04074473
Title: Impact of Nonselective Beta-blocker on Acute Kidney Injury in Cirrhotic Patients With Esophageal Varices
Acronym: AKI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-04-014A
Record Dates: First submitted 2019-08-29; First posted 2019-08-30 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Acute Kidney Injury; Cirrhosis; Esophageal Varices
Keywords: portal hypertension, esophageal varices, non-selective beta-blocker, acute kidney injury.
MeSH Terms: conditions — Acute Kidney Injury; Fibrosis; Esophageal and Gastric Varices; Hypertension, Portal | interventions — Propranolol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Propranolol alone (Placebo Comparator): TPropranolol 10mg BID initially and titrate dosage every week to achieve 25% drop of heart rate (keep heart rate>55 or systemic blood pressure>90mmHg)
  Interventions: Drug: propranolol
- Esophageal variceal ligation alone (Active Comparator): Esophageal variceal ligation every 3-4 weeks to achieve variceal eradication under endoscopy. After eradication, follow-up endoscopy every 3 months and variceal ligation again if recurrence.
  Interventions: Procedure: Esophageal varice ligation
- Esophageal variceal ligation(DC inderal after EV eradication) (Experimental): Patients randomized to banding ligation group discontinue propranolol after eradication of esophageal varices.
  Interventions: Other: DC propranolol
- Propranolol(Keep BB after EV eradication) (No Intervention): Patients randomized to propranolol group continue propranolol after eradication of esophageal varices.

INTERVENTIONS:
Drug: propranolol — Propranolol 10mg BID initially and titrate dosage every week to achieve 25% drop of heart rate (keep heart rate>55 or systemic blood pressure>90mmHg)
  Arms: Propranolol alone
Procedure: Esophageal varice ligation — Esophageal variceal ligation every 3-4 weeks to achieve variceal eradication under endoscopy
  Arms: Esophageal variceal ligation alone
Other: DC propranolol — Patients randomized to banding ligation group discontinue propranolol after eradication of esophageal varices.
  Arms: Esophageal variceal ligation(DC inderal after EV eradication)

SUMMARY:
We will include patients with EV and EVB. They will be randomized to EVL vs. NSBB for primary prevention And EVL+long-term NSBB vs. EVL+short-term NSBB for secondary prevention. 150 patients will be included in a 3-year period. Primary end-points are formation/progression of ascites, acute kidney injury and survival. The other outcomes such as bleeding, rebleeding, infection and other risk factors will be also analyzed.

DETAILED DESCRIPTION:
Despite advance in the prevention and treatment of esophageal variceal bleeding (EVB), it is still a majorcomplication of portal hypertension with the characteristic of a high mortality around 15~20% after anepisode of hemorrhage. Following development of EV and EVB, ascites and renal dysfunction occurs in a large portion of patients with time. The international consensus suggested use of non-selective beta-blocker(NSBB) to prevent EVB. Long-term use of NSBB was also found to decrease occurrence of encephalopathy and spontaneous bacterial peritonitis (SBP) and extend survival. Until 2010, Dr. Lebrec et al. found use of NSBB might decrease survival in cirrhotic patients with refractory ascites, therefore they suggested discontinued use of NSBB in these patients. The findings lead to a vigorous dispute between hepatologists. In 2011, the reputable team again found use of NSBB might cause post-paracentesis circulatory dysfunction (PPCD) in cirrhotic patients undergoing a large volume paracentesis. Occurrence of PPCD was known to cause acute kidney injury (AKI) and increase mortality. In 2014, Austria investigators found use of NSBB was associated with increased AKI and shortened survival in patients with SBP. Despite the findings of these studies implicated the harmful aspects of NSBB use, a major debate remained because lack of randomized controlled trial some unequal distribution of patients.Taipei Veterans General Hospital is renowned by its high profile research in portal hypertension and its related complications. The current proposal is aimed to clarify the strategy of NSBB use. We will include patients with EV and EVB. They will be randomized to EVL vs. NSBB for primary prevention And EVL+long-term NSBB vs. EVL+short-term NSBB for secondary prevention. 150 patients will be included in a 3-year period. Primary end-points are formation/progression of ascites, acute kidney injury and survival. The other outcomes such as bleeding, rebleeding, infection and other risk factors will be also analyzed.

ELIGIBILITY:
Criteria

Inclusion Criteria:

Age of 20 to 85 years

Cirrhotic patients with esophageal varices regardless of bleeding event or not will be enrolled in this study.

Exclusion Criteria:

Terminal stage HCC/ other malignancy/ Stroke or active sepsis/ Chronic kidney disease stage 4 under renal replacement therapy/ Contraindications to non-selective beta-blockers/ A history of non-selective beta-blockers use, sclerotherapy, banding ligation, transjugular intrahepatic porto-systemic shunt, or shunt surgery/ Serum total bilirubin >10 mg/dL/ Refractory ascites/ Hepato-renal syndrome/ Pregnancy/ Severe heart failure (NYHA Fc III/IV)/ Bronchial asthma or chronic obstructive pulmonary disease/ Second or third degree atrioventricular block/ Severe hypotension/ Refusal to participate

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2015-04-13; Primary Completion 2015-11-05 (Actual); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Acute kidney injury | 3 years
Heparenal syndrome | 3 years
overall survival | 3 years

SECONDARY OUTCOMES:
EV bleeding/rebleeding | 3 years
Infection rate | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan